CLINICAL TRIAL: NCT05256199
Title: Dutch Multidomain Lifestyle Intervention in Older Adults at Risk of Cognitive Decline
Acronym: FINGER-NL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alzheimercentrum Amsterdam (Other)
Collaborators: Maastricht University (Other); Radboud University Medical Center (Other); Wageningen University and Research (Other); University Medical Center Groningen (Other); Danone Nutricia Research (Industry)
Responsible Party: Principal Investigator, Marissa Zwan, ass. PI, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021.0220; NL77242.029.21 (Other: Centrale Commissie Mensgebonden Onderzoek (CCMO))
Record Dates: First submitted 2022-01-11; First posted 2022-02-25 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Cognitive Decline; Life Style; Risk Reduction
MeSH Terms: conditions — Cognitive Dysfunction; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-intensity group (Experimental): The high intensity group receives a personalized, supervised intervention consisting of group meetings and individual sessions.
  Interventions: Behavioral: Multidomain lifestyle intervention
- low-intensity group (No Intervention): The low-intensity arm receives online access to general lifestyle-related health information.

INTERVENTIONS:
Behavioral: Multidomain lifestyle intervention — A multidomain lifestyle intervention, including (1) physical activity, (2) cognitive training, (3) cardiovascular risk factor management (Cardiovascular), (4) dietary counselling, (5) Souvenaid, (6) sleep counselling, (7) stress management, and (8) social activities.
  Arms: high-intensity group

SUMMARY:
FINGER-NL is a multi-center, randomized, controlled, multidomain lifestyle intervention trial among 1,206 older adults at risk for cognitive decline with a duration of 24 months. Participants are randomized in a 1:1 ratio to a personalized multi-domain lifestyle intervention (high-intensity intervention group) versus online access to general lifestyle-related health information (low-intensity intervention group). After the intervention period, participants are invited for a 24 month extension of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 60-79 years of age at pre-screening;
* Adequate fluency in Dutch to understand the informed consent and complete questionnaires;
* Providing informed consent to all study procedures;
* Internet access at home;
* Presence of ≥3 self-reported risk factors for cognitive decline (must contain at least 2 modifiable risk factors and 1 non-modifiable riskfactor).

Exclusion Criteria:

* Diagnosis of dementia or mild cognitive impairment at baseline (self-reported);
* Significant cognitive impairment assessed using the Modified Telephone Interview for Cognitive Status battery (TICSm score<23);
* Conditions affecting safe and continuous engagement in the intervention (e.g. under treatment for current malignant diseases, major psychiatric disorders (e.g. major depression, psychosis, bipolar disorder), neurological disorders (e.g. Parkinson's disease, multiple sclerosis), symptomatic cardiovascular disease (e.g. stroke, angina pectoris, heart failure, myocardial infarction), re-vascularization within three months, severe loss of vision, hearing or communicative ability, severe mobility impairment, other conditions preventing co-operation) as judged by the local study nurse or consulted physician at the local study site;
* Coincident participation in any other intervention trial at time of pre-screening.
* Coincident participation of spouse in FINGER-NL trial.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1210 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
2-year change from baseline in global cognitive composite score | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Global cognitive composite score derived from subtest scores from the Neuropsychological Test Battery (NTB) that includes 15-Word Verbal Learning Test delayed recall (discrete number; 0-15 (higher score means a better outcome)), Digit Symbol Substitution Test 90 seconds (discrete number; 0-90 (higher score means a better outcome)), WAIS digit span backwards (discrete number; 0-14 (higher score means a better outcome)), and semantic fluency (discrete number; 0-no maximum, higher score means a better outcome)).

SECONDARY OUTCOMES:
15-Word Verbal Learning Test delayed recall | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  discrete number; score: 0-15 (higher score means a better outcome)
Digit Symbol Substitution Test 90 seconds | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  discrete number; 0-90 (higher score means a better outcome)
Wechsler Adult Intelligence Scale (WAIS) digit span backwards | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  discrete number; 0-14 (higher score means a better outcome)
Semantic fluency | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  word count in one minute; minimum 0, no maximum, higher score means a better outcome.
Instrumental activities of daily living using the Amsterdam Instrumental Activity of Daily Living Questionnaire (A-IADL-Q) | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Total scores range approximately 20-70, higher scores indicate better IADL functioning
5 level EuroQol-5D (EQ-5D-5L) | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Quality of life, score 0-100, higher scores indicate better quality of life
LIfestyle for BRAin health (LIBRA) | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Modifiable dementia risk using lifestyle for brain health; The score ranges from -5.9 (minimum score) to +12.7 (maximum score), with higher scores meaning a worse outcome (higher dementia risk)
grip strength test | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Scores between 0 to 90 kg can be measured on the Jamar Hand dynamometer, with higher scores indicating better grip strength
SQUASH questionnaire | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  METs derived from the Ainsworth's compendium of physical activity will be used to classify physical activity intensity (<1.5METs- sedentary, 1.6-2.9 METs- light, 3.0-5.9METs- moderate, >6.0- vigorous physical activity).
LASA Sedentary Behavior Questionnaire | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Average hours and minutes of sedentary behavior a day, range from 0 to 24 hours. Higher scores (more hours) means a more sedentary behavior.
Pittsburgh Fatigability Scale | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Total physical and mental fatigability scores range from 0-50, with higher scores indicating higher fatigability.
SARC-F Sarcopenia Questionnaire | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  sarcopenia, scores range from 0 to 10 (i.e. 0-2 points for each component; 0 = best to 10 = worst).
Five Facet Mindfulness Questionnaire - Short Form (FFMQ-SF) | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Total scale ranges from 24 - 120, higher scores indicate more mindfulness
Perceived Stress Scale | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Total score, scale 0 - 40, higher scores indicate more perceived stress
MetaMemory in Adulthood (MIA) | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Sum of Part 1 + Part 2A and B. Part 1: Strategy (scores 10 - 50, higher scores indicate more use of strategies), Part 2A: Subjective memory functioning, scores ranges from 23 - 115, with higher scores indicate better memory self-efficacy and 2B: Locus, scores ranges from 7 - 35, higher scores indicate better perceived personal control over remembering abilities.
Blood pressure | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  scores range from approximately (for diastolic) 60-120 and (for systolic) 100-180 mmHg, with higher scores indicating higher blood pressure.
Cholesterol | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  total (healthy level: 125 to 200mg/dL), HDL (healthy level = 40mg/dL or higher), LDL (healthy level = Less than 100mg/dL) + triglycerides (healthy level = less than 150-199 mg/dL)
Blood glucose | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  HbA1C, scores range from approximately 30-100 mmol/mol, with higher scores indicate higher blood glucose levels.
Waist circumference | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  measured in cm
Hip circumference | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  measured in cm
Height | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  measured in cm
Weight | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  measured in kg
Hill-Bone Medication Adherence Scale | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  scores range from 9-26, with lower scores indicating better medication adherence
MIND-adjusted Eetscore-FFQ | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Dutch Healthy Diet Index 2015 score (range 0-160 points, higher scores mean better outcome) and MIND score (range 0-15 points, higher scores mean better outcome), assessed by a short Food Frequency Questionnaire.
Nutritional intake | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Change in nutritional intake measured by an online 3-day food diary (assessed by Traqq application), qualitative assessment
Pittsburg Sleep Quality Index | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  Total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality
Insomnia severity index | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  The score ranges from 0 (minimum score) to 28 (maximum score), with lower scores indicating a better outcome
Lubben Social Network Scale | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  The score ranges from 0 (minimum score) to 30 (maximum score), with higher scores meaning a better outcome (higher level of perceived social support)
De Jong Gierveldt Loneliness Scale | 2 years (measured at baseline and follow-up 2)
  The score ranges from 0 (minimum score) to 6 (maximum score), with higher scores representing a worse outcome (higher loneliness scores)
Aβ42/40 ratio | 2 years (measured at baseline and follow-up 2)
  amyloid-β (1-42)/(1-40) (pg/mL)
p-tau | 2 years (measured at baseline and follow-up 2)
  phosphorylated tau (pg/mL)
NfL | 2 years (measured at baseline and follow-up 2)
  neurofilament light chain (pg/mL)
GFAP | 2 years (measured at baseline and follow-up 2)
  glial fibrillary acidic protein (pg/mL)
BDNF | 2 years (measured at baseline and follow-up 2)
  brain-derived neurotrophic factor (pg/mL)
Actigraph (Groningen site only) | 2 year (measured for 1 week at baseline, follow-up 1 and follow-up 2)
  physical activity, sedentary behavior and sleep-wake activity
Physical Activity Record questionnaire (Groningen site only) | 2 year (measured for 1 week at baseline, follow-up 1 and follow-up 2)
  physical activity, sedentary behavior and sleep-wake activity

OTHER OUTCOMES:
MOCA | baseline
  Montreal Cognitive Assessment, minimum score 0, maximum score 30, with higher scores indicating better cognitive performance
Motivation to Change Lifestyle and Health Behavior for Dementia Risk Reduction scale | 2 years (measured at baseline, follow-up 1 and follow-up 2)
  scores range from 27-135, with higher scores indicating greater motivation to change

CONTACTS AND LOCATIONS:
Overall Officials: Wiesje M van der Flier, Prof, Principal Investigator — Alzheimer Center Amsterdam; Sebastian Köhler, Ass Prof, Principal Investigator — Maastricht University
Locations (5):
- Netherlands (5):
  - Alzheimer Center Amsterdam, Amsterdam
  - University Medical Center Groningen, Groningen
  - Maastricht University, Maastricht
  - Radboud University, Nijmegen
  - Wageningen Unversity and Research, Wageningen

REFERENCES:
- [Derived] Deckers K, Zwan MD, Soons LM, Waterink L, Beers S, van Houdt S, Stiensma B, Kwant JZ, Wimmers SCPM, Heutz RAM, Claassen JAHR, Oosterman JM, de Heus RAA, van de Rest O, Vermeiren Y, Voshaar RCO, Smidt N, Broersen LM, Sikkes SAM, Aarts E; MOCIA consortium; FINGER-NL consortium; Kohler S, van der Flier WM. A multidomain lifestyle intervention to maintain optimal cognitive functioning in Dutch older adults-study design and baseline characteristics of the FINGER-NL randomized controlled trial. Alzheimers Res Ther. 2024 Jun 13;16(1):126. doi: 10.1186/s13195-024-01495-8. PMID 38872204